CLINICAL TRIAL: NCT06998680
Title: A 6-Month Randomized Double-Blind Placebo-Controlled Trial Assessing the Efficacy of Oral and Topical Traditional Chinese Medicine Products on Alopecia and Canities
Brief Title: 6-Month Trial of Chinese Herbal Treatments for Hair Loss and Gray Hair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vita Green Pharmaceutical (H.K.) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025011301
Record Dates: First submitted 2025-04-17; First posted 2025-05-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-05

CONDITIONS: Alopecia; Canities
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VitaGreen Capsule A+VitaGreen Tonic (Experimental)
  Interventions: Other: VitaGreen Capsule A+VitaGreen Tonic
- VitaGreen Capsule B+VitaGreen Tonic (Experimental)
  Interventions: Other: VitaGreen Capsule B+VitaGreen Tonic
- Capsule Placebo+VitaGreen Tonic (Experimental)
  Interventions: Other: Capsule Placebo+VitaGreen Tonic
- Capsule Placebo+Tonic Placebo (Placebo Comparator)
  Interventions: Other: Capsule Placebo+Tonic Placebo

INTERVENTIONS:
Other: VitaGreen Capsule A+VitaGreen Tonic — VitaGreen Capsule A+VitaGreen Tonic,use 24 weeks
  Arms: VitaGreen Capsule A+VitaGreen Tonic
Other: VitaGreen Capsule B+VitaGreen Tonic — VitaGreen Capsule B+VitaGreen Tonic,use 24 weeks
  Arms: VitaGreen Capsule B+VitaGreen Tonic
Other: Capsule Placebo+VitaGreen Tonic — Capsule Placebo+VitaGreen Tonic,use 24 weeks
  Arms: Capsule Placebo+VitaGreen Tonic
Other: Capsule Placebo+Tonic Placebo — Capsule Placebo+Tonic Placebo,use 24 weeks
  Arms: Capsule Placebo+Tonic Placebo

SUMMARY:
This will be a 6-month randomized, double-blind, placebo-controlled trial. A total of 152 participants with hair loss, including some with gray hair, will be enrolled and randomly assigned to four groups. Each group will receive a combination of oral capsules and hair tonic, to be used as directed for 24 weeks. Participants will attend three in-person visits, during which assessments-including hair-related tests and photographs-will be conducted to evaluate hair count and density. Additionally, 10 participants with gray hair from each group will undergo extra assessments focused on changes in hair color. All relevant clinical data will be systematically collected and recorded for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign the informed consent form prior to enrollment and fully understand the study's purpose, procedures, and potential adverse events.
2. Adults aged 18 to 60 years, both male and female; each group must include no less than 50% female participants.
3. Hair length must be greater than 5 cm.
4. Women must meet the Savin scale classification between grades 1-3 to II.
5. Men must meet the Norwood-Hamilton classification between stages II and VI.
6. At least 10 participants in each group must have gray hair, with a minimum of 5 gray hairs within a 1 cm × 4 cm area of the scalp.
7. Participants must not have undergone any special hair treatments-such as dyeing, perming, or styling-within the past two months.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or individuals planning to conceive in the near future.
2. Individuals with medical conditions causing hair loss, such as refractory alopecia areata, inflammatory scarring alopecia, or psoriatic alopecia; or those diagnosed with other scalp or hair disorders.
3. Individuals with diagnosed psychiatric or psychological disorders, or those with long-term sleep disturbances or emotional regulation issues.
4. Use of anti-hair loss cosmetics or other hair growth-promoting products within the past 3 months.
5. Use of any systemic or topical medications known to affect hair growth within the past 6 months.
6. History of hair transplantation.
7. Curly hair.
8. Individuals with highly sensitive constitutions.
9. Individuals diagnosed with severe anemia or abnormal liver/kidney function during physical examination.
10. Participation in any other clinical trials involving the test area within the past 2 months.
11. Any other conditions deemed unsuitable for participation by the clinical investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Hair Shedding Count | Baseline, week 12, week 24
  Combing the hair 60 times and recording the number of hairs that fall out during the process
Local Hair Count | Baseline, week 12, week 24
  Detected by Dermatoscope
Local Hair Density | Baseline, week 12, week 24
  Detected by Dermatoscope
percentage of Vellus Hair | Baseline, week 12, week 24
  Detected by Dermatoscope
Percentage of Terminal Hair | Baseline, week 12, week 24
  Detected by Dermatoscope
Scoring of Hair Changes from Images | Baseline, week 12, week 24
  Doctor scores hair changes from Images pictured by camera with scale of 0 to 4

SECONDARY OUTCOMES:
local hair color scores and white hair Index | Baseline, week 12, week 24
  Doctor evaluates local hair color scles according to Wig Color Grading（Value1 to Value 6）and calculates the white hair Index
Complete Blood Count concentrations | Baseline, week 24
  Blood sample detected by Hematology Analyzer
Urinalysis concentrations | Baseline, week 24
  Urine sample detected by Urine Analyzer
Aspartate Aminotransferase concentrations | Baseline, week 24
  Blood sample detected by Biochemical analyzer
Alanine Aminotransferase concentrations | Baseline, week 24
  Blood sample detected by Biochemical analyzer
Creatinine concentrations | Baseline, week 24
  Blood sample detected by Biochemical Analyzer
Urea Nitrogen concentrations | Baseline, week 24
  Blood sample detected by Biochemical Analyzer
Serum Uric Acid concentrations | Baseline, week 24
  Blood sample detected by Biochemical Analyzer
Adverse Events | Baseline, week 24
  counting and documenting adverse events happening during the experiment

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Xiangtan City, Xiangtan, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes